CLINICAL TRIAL: NCT07064512
Title: The Effect of Exertional and Exogenous Heating on Physiological Markers
Brief Title: The Effect of Heat Exposure on Physiological Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian Sports University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: LithuananianSportsU-24
Record Dates: First submitted 2025-07-11; First posted 2025-07-14 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Healthy Adult Male

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exogenous heating (Experimental): Healthy young subjects participated received exogenous heating modality, where the participants sat immersed in a water bath at 43.5 ± 0.5°C and remained submerged until rectal temperature reached 39°C.
  Interventions: Other: Exogenous heating
- Endogenous heating (Experimental): Healthy young subjects participated received endogenous heating modality, the participant cycled at 60% of his VO2max until rectal temperature reached 39°C
  Interventions: Other: Endogenous heating

INTERVENTIONS:
Other: Endogenous heating — Exercise was used as the endogenous heating modality, the participant cycled at 60% of his VO2max until rectal temperature reached 39°C
  Arms: Endogenous heating
Other: Exogenous heating — Hot-water immersion was used as the exogenous heating modality, where the participants sat immersed in a water bath at 43.5 ± 0.5°C and remained submerged until rectal temperature reached 39°C.
  Arms: Exogenous heating

SUMMARY:
This study is the first to examine the effects of core temperature elevation on kynurenine pathway (KP) metabolites in healthy young males. It was hypothesized that rise in core temperature due to both pasive heating and exercise will initiate a stress response, affecting the concentration of KP metabolites. Additionally, it was expected that the exercise would produce more pronounced effects due to the increased cardiovascular, mechanical, and metabolic demands associated with it. Thus, the the main purpose of the present study was to investigate and to compare the effects of two distinct heat stress modalities on KP metabolites.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults;
* age between 18 - 36 years;
* physically active (exercising 2-3 times per week);
* non-smoking.

Exclusion Criteria:

* a body mass index (BMI) > 30 kg/m2;
* neurological, cardiovascular, metabolic, and/or inflammatory diseases, or conditions that could be worsened by exposure to interventions and that could affect experimental variables;
* involvement in temperature manipulation program for ≥ 3 months.

Ages: 18 Years to 36 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
Change in plasma metabolites of the kynurenine pathway (μm) | Day 1 (every 0.5 °C until rectal temperature (Trec) reached 39°C, followed by a recovery phase until Trec reached 37.5°C)
  An ultra-performance liquid chromatography-tandem mass spectrometry system (UPLC-MS/MS) was used to measure venous plasma levels of tryptophan, kynurenine, kynurenic acid, 3-hydroxy-kynurenine, quinolinic acid, nicotinamide and picolinic acid (in μm). The UPLC-MS/MS system uses a Xevo TQ-XS triple quadrupole mass spectrometer (Waters) with a Z-spray electrospray interface, and the system operates in electrospray positive multiple reaction monitoring mode.
Rectal temperature (°C) | Day 1 (during both heating modalities until Tre reached 39°C, followed by a recovery phase until Trec reached 37.5°C)
  Rectal temperature (in °C) was measured using a thermocouple (Rectal Probe, Ellab, Denmark) inserted to a depth of 12 cm past the anal sphincter.
Change in heart rate (bpm) | Day 1 (during both heating modalities until Tre reached 39°C, followed by a recovery phase until Trec reached 37.5°C)
  Heart rate (in bpm) was recorded using a heart rate sensor with a chest strap (Polar, Finland).
Change in physiological strain index | Day 1 (every 0.5 °C until rectal temperature (Trec) reached 39°C, followed by a recovery phase until Trec reached 37.5°C)
  A physiological strain index (PSI) was used to indicate heat strain. PSI = 5 x (Tret - Tre0) x (39.5 - Tre0)^-1+ 5 x (HRt - HR0) x (180 - HR0)^-1, where rectal temperature (Tre) t and heart rate (HR) t are simultaneous measurements taken every 0.5°C of the heat exposure and Tre0 and HR0 are the initial measurements.
Change in glucose (mmol/L) | Day 1 (every 0.5 °C until rectal temperature (Trec) reached 39°C, followed by a recovery phase until Trec reached 37.5°C)
  The glucose concentration (in mmol/L) was measured using an automatic blood glucose meter Glucocard X-mini-Plus (Arkray Inc, Japan).
Change in lactate (mmol/L) | Day 1 (every 0.5 °C until rectal temperature (Trec) reached 39°C, followed by a recovery phase until Trec reached 37.5°C)
  The lactate concentration (in mmol/L) was measured using an Accutrend Plus System (Roche, Germany).
Changes in prolactin concentration (ng/mL) | Day 1 (every 0.5 °C until rectal temperature (Trec) reached 39°C, followed by a recovery phase until Trec reached 37.5°C)
  The venous prolactin (in ng/mL) was measured using enzyme-linked immunosorbent assay kit and a Spark multimode microplate reader (Tecan, Austria).
Changes in catecholamines concentration (ng/mL) | Day 1 (every 0.5 °C until rectal temperature (Trec) reached 39°C, followed by a recovery phase until Trec reached 37.5°C)
  The venous adrenaline and noradrenaline concentrations (in ng/mL) was measured using enzyme-linked immunosorbent assay kits and a Spark multimode microplate reader (Tecan, Austria).
Changes in salivary cortisol concentration (µg/dL) | Day 1 (every 0.5 °C until rectal temperature (Trec) reached 39°C, followed by a recovery phase until Trec reached 37.5°C)
  The saliva samples was collected to measure cortisol level (in µg/dL) using an ELISA kits and a Spark multimode microplate reader (Tecan, Austria).

CONTACTS AND LOCATIONS:
Locations (1):
- Lithuanian Sports University, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided